CLINICAL TRIAL: NCT04697329
Title: Laparoscopic Cholecystectomy: Use of Infiltration With Levobupivacaine and Postoperative Pain: A Randomized Controlled Trial
Brief Title: Local Infiltration With Levobupivacaine During Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Móstoles (Other)
Responsible Party: Principal Investigator, JORGE HERRADOR BENITO, Principal Investigator. Surgeon., Hospital Universitario de Móstoles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUMOSDEC2020
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Pain; Local Infiltration; Levobupivacaine
Keywords: Laparoscopic cholecystectomy; Postoperative Pain; Local Infiltration; Levobupivacaine; Randomized controlled trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local infiltration (Experimental)
  Interventions: Drug: Preincisional infiltration with levobupivacaine
- No local infiltration (No Intervention)

INTERVENTIONS:
Drug: Preincisional infiltration with levobupivacaine — Local, preincisional infiltration of port sites with levobupivacaine 5 mg/ml 20 ml
  Arms: Local infiltration

SUMMARY:
Randomized controlled trial on laparoscopic cholecystectomy. Interventional group: preincisional infiltration with levobupivacaine. Control group: no local infiltration.

Postoperative pain with numeric rating scale is registered, besides other parameters like heart rate, blood pressure, rescue analgesia requirements, nausea and vomiting, etc.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patient refusal
* Open surgery
* Reintervention surgery
* Drain tube placement
* Cognitive impairment
* Allergic reactions to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessed by visual numeric scale. | 24 hours
  Values come from 0 to 10, where 0 means no pain and 10 means the worst imaginable pain. Best outcome would be 0 or close to 0

SECONDARY OUTCOMES:
Postoperative administration of analgesics | 24 hours
  Record of dose of analgesics needed: nonsteroidal anti-inflamatory drugs, opioid requirements, other analgesics requirements
Postoperative nausea and vomiting episodes | 24 hours
  Record of episodes of nausea or vomiting during first 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL DURÁN POVEDA, MD, Study Director — H. U. REY JUAN CARLOS; GIL RODRÍGUEZ CARAVACA, MD, Study Director — H. F. ALCORCÓN
Locations (1):
- Hospital Universitario de Móstoles, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: March 2022. 6 months.